CLINICAL TRIAL: NCT06048835
Title: Ultrasensitive BIOsensing Platform for Multiplex CELLular Protein PHEnotyping at Single-cell Level
Brief Title: Circulating Tumour Cells Characterization in Breast Cancer Patients
Acronym: BioCellPhe
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Carlo Morasso (Unknown)
Responsible Party: Principal Investigator, Fabio Corsi, Professor, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2684
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MBC: Patients diagnosed with metastatic breast cancer
  Interventions: Device: Blood sample
- EBC: Patients diagnosed with primary early-breast cancer candidate for surgery
  Interventions: Device: Blood sample
- HC: Control group of sex and age matched healthy volunteers, not affected by any neoplastic disease
  Interventions: Device: Blood sample

INTERVENTIONS:
Device: Blood sample — For each patient, a 15 ml EDTA blood sample will be collected at different time-points

SUMMARY:
In the current scenario, a reliable liquid biopsy method for predicting outcomes in solid tumors, especially among breast cancer patients, is lacking. Circulating Tumor Cells (CTCs) serve as crucial indicators of metastasis, and their early detection could significantly enhance patient stratification and facilitate the customization of personalized treatments. However, detecting CTCs in breast cancer patients presents complexities due to their substantial phenotypic heterogeneity and typically low concentration.

Numerous approaches have been developed for CTC detection. Nonetheless, the currently available technologies remain intricate, time-consuming, and costly. The BioCellPhe Project is dedicated to the development of a novel device capable of isolating and characterizing individual CTCs. This innovative device relies on the identification of specific cell membrane proteins with remarkable precision, achieved through the application of novel orthogonal techniques.

On one hand, engineered bacteria are utilized to precisely bind to membrane proteins of interest on CTCs. On the other hand, Surface Enhanced Raman Spectroscopy (SERS) is employed for the detection of individual molecules. Specifically, the BioCellPhe Project focuses on comprehensively studying CTCs in breast cancer patients, encompassing both metastatic and non-metastatic cases.

DETAILED DESCRIPTION:
This is an experimental, prospective and monocentric study. This study involves consecutive patients with diagnosis of breast cancer (BC), including early breast cancer and metastatic breast cancer patients, referring to the Breast Unit and to the Oncology Department at Istituti Clinici Scientifici Maugeri, Pavia (Italy).

Patients diagnosed with different histological types of breast cancer will be enrolled in the study: luminal BC, HER2-enriched BC, triple-negative BC.

The study duration is 24 months, starting from December 2022 to December 2024.

The patients will be divided into three groups, as follows:

* Population 1: patients diagnosed with metastatic breast cancer.
* Population 2: patients diagnosed with primary early-breast cancer candidate for surgery.
* Population 3: a control group of sex and age matched healthy volunteers, not affected by any neoplastic disease.

For each patient, a 15 ml EDTA blood sample will be collected at different time-points, as follows:

* Population 1: before starting a potential chemotherapy treatment.
* Population 2: before undergoing surgical procedure.
* Population 3: at the first useful moment. The blood samples will be collected at the Maugeri Institute and CTCs will be isolated within 48 hours to validate the device.

For each patient, the following clinico-anamnestic information will be collected: age, histological tumour information at diagnosis (tumour subtype, grading, receptors' status, Ki-67 value), histological metastases information, clinical stage (clinical TNM), type of surgery, pathological staging after surgery (pTNM).

ELIGIBILITY:
Inclusion Criteria:

* female patients with diagnosis of metastatic breast cancer, confirmed by clinical practice staging exams.
* female patients with biopsy-confirmed diagnosis of early-breast cancer candidate for primary surgery after multidisciplinary evaluation.
* patients not affected by any neoplastic disease.

Exclusion Criteria:

* Diagnosis of any neoplastic disease

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is referred to women
Study Population: The study involves female patients with diagnosis of early-breast cancer candidate for surgery and female patients with diagnosis of metastatic breast cancer. A control group of sex and age matched healthy volunteers, not affected by any neoplastic disease will be enrolled too.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detect specific proteins on CTCs in breast cancer patients | 24 months
  Clinical validation of a new technological device able to detect specific target surface proteins on CTCs in breast cancer patients, both non-metastatic and metastatic.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No